CLINICAL TRIAL: NCT06633705
Title: Investigation of the Effects of Local Estrogen Administration on Vaginal, Periurethral and Urinary Microbiota in Genitourinary Syndrome
Brief Title: Changes in Neighbouring Microbiota in Genitourinary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Koc University Hospital (Other)
Responsible Party: Principal Investigator, Sebile Guler Cekic, MD-PhD, Koc University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023.049.IRB1.012
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: Genitourinary Syndrome of Menopause; vaginal microbiota; periurethral microbiota; urobiome
MeSH Terms: interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: There are 2 intervention groups and 2 control groups. Control group1 consists of menopause patients without symptoms of GUS and examination findings. Control group 2 consists of menopause patients without symptoms of GUS but have examination findings.
  Intervention groups are those with GUS symptoms. They were randomly divided in 2 groups: one group had vaginal oestrogen treatment first other group had the treatment after the samples were taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GUS-estriol (Experimental): Patients with GUS symptoms and examination findings, who are treated with vaginal oestrogen cream
  Interventions: Drug: Vaginal Cream with Applicator
- GUS-control (No Intervention): Patients with GUS symptoms and examination findings
- Control M (No Intervention): Patients in menopause who doesn't have any GUS symptoms nor examination findings
- Control AV (No Intervention): Patients in menopause who doesn't have any GUS symptoms but have examination findings

INTERVENTIONS:
Drug: Vaginal Cream with Applicator — Vaginal Cream that contains estriol (1mg estriol in 1 g cream)
  Arms: GUS-estriol

SUMMARY:
Genitourinary syndrome (GUS) is a disease seen in menopause, which significantly reduces the quality of life of patients. Microbiota studies in GUS are mostly related to vaginal microbiota. However, although urinary problems are also common in GUS, there are less studies on urobiome and no studies on periurethral microbiota. It is recently shown that especially in patients with dyspareunia vaginal microbiota mostly consists of Streptococcus species. As periurethral tissues are close to the skin it is reasonable to think that periurethra and vaginal opening may be colonised by aerobic bacteria which causes the symptoms like burning sensation and dyspareunia. The hypothesis of the study is that vaginal dysbiosis and related aerobic bacteria that become dominant in the periurethral microbiota may be responsible for the emergence of symptoms in menopausal patients with genitourinary syndrome. Changes in the vaginal microbiota with vaginal estrogen therapy will lead to changes in the urobiome and periurethral microbiota. Our aim is to determine the vaginal, periurethral and urinary microbiota content of menopausal women with genitourinary syndrome, to determine the effect of local estrogen therapy on them, and to examine whether there is a difference between these 3 microbiota.

DETAILED DESCRIPTION:
Problems addressed by the study:

Genitourinary syndrome (GUS) is a common disorder during menopause, reported to be at least 50% in many series, which reduces quality of life. Unfortunately, despite being such a common disorder, patients do not report their complaints about this issue and clinicians do not question patients about this condition (NAMS, 2020). There is little awareness about the subject and relatively few studies on the pathophysiology and treatment of the disease.

GUS is diagnosed clinically. Symptoms such as vulvovaginal dryness, burning or irritation; dyspareunia; and symptoms such as urge incontinence, dysuria or recurrent urinary tract infections are observed in the urinary system (NAMS, 2020). Urinary symptoms of GUS, such as dysuria, are often confused with recurrent urinary tract infections. The pathophysiology of GUS is often attributed to estrogen deficiency, but some researchers suggest that these changes may also be related to the vaginal microbiome (Hummelen et al., 2011). Because while estrogen deficiency is present in all women who enter menopause, GUS is observed in a certain portion. Therefore, our study will contribute to the literature aimed at shedding light on the pathogenesis.

Although there are both vaginal and urinary symptoms in GUS, the most studies are on vaginal microbiota. There is only one study on urinary microbiota (Lillemon et al., 2022). There is no study evaluating the periurethral microbiota.

Is there a relationship between vaginal microbiota and GUS symptoms?

The relationship between vaginal microbiota and GUS has been addressed in many studies. Various changes occur in the vaginal flora during menopause due to the decrease in estrogen hormone during menopause. Gustafsson et al. (2011) reported that women of reproductive age were more frequently colonized with L. crispatus compared to menopausal women. Similarly, premenopausal women had significantly higher free glycogen levels and higher Lactobacillus levels compared to postmenopausal women (Zhang et al., 2012; Mirmonsef et al., 2014).

Studies on patients with GUS symptoms have shown that women with mild GUS symptoms were more likely to be predominantly Lactobacillus species in the vagina and had lower bacterial diversity, whereas in more severe GUS cases, colonization with Lactobacillus species was reduced and there was greater bacterial diversity (Brotman et al., 2018). Species detected in the group with increased bacterial diversity included Prevotella, Porphyromonas, Peptoniphilus and Bacillus (Brotman et al., 2018). Notably, CST IV-A colonization was more prevalent in the vagina in women with the most severe GUS symptoms (Hummelen et al., 2011, Brotman et al., 2018).

In the studies summarized here, a vaginal microbiota dominated by Lactobacillus species was detected in all women receiving hormone replacement therapy or local estrogen therapy, suggesting that estrogen levels have an effect on the vaginal bacterial community and structure. However, whether GUS symptoms are reduced by estrogen-related changes or by changes in the vaginal flora is still controversial. Although many studies have shown that Lactobacillus dominance in the vaginal microbiota is negatively associated with GUS symptoms, studies have recently been published showing that this is not the case. Mitchell compared 3 groups given local estrogen, vaginal lubricant, and placebo in their study (Mitchell, 2018). GUS complaints decreased in all three of these groups; vaginal estradiol -1.4 (95%CI, -1.6 to -1.2); moisturizer, -1.2 (95%CI, -1.4 to -1.0); and placebo, -1.3 (95%CI, -1.5 to -1.1). Although the amount of Lactobacilli increased significantly in the local estrogen group compared to the other groups, the similar decrease in complaints cannot be explained by both estrogen and microbiota hypotheses.

We planned to use 2 different control groups in our study to investigate this issue. Patients without any GUS symptoms and without vulvovaginal atrophy findings on examination will be the first control group, and patients without complaints but with vulvovaginal atrophy findings on examination will be the second control group. Examining whether there is a difference in colonization in these two groups will be the first in the literature and will contribute to the literature in terms of elucidating the pathogenesis.

As mentioned before there are both vaginal and urinary symptoms in GUS. So is there a relationship between vaginal microbiota and periurethral and urinary microbiota? There is a study on this subject that examined both vaginal and urinary microbiota. In the study, local estrogen treatment neither caused a significant decrease in GUS symptoms nor caused a change in vaginal and urinary microbiota (Lillemon et al., 2022). In this study, Lillemon and his team examined the effect of local estrogen treatment on vaginal and urinary microbiota separately and did not examine whether there were similarities or differences between the two environments. In addition, since they included patients who were generally in menopause and not those with only GUS complaints in the study, local estrogen treatment was found to be unsuccessful. Yet, local estrogen treatment is the first-line treatment after lubricants in GUS and is a successful treatment method in 85% of patients (NAMS, 2020). Since they used a general menopausal population in the study, there may not have been a significant difference in microbiota between patients taking estrogen and those not taking it, and a significant decrease in GUS complaints in those taking local estrogen.

There is no study comparing vaginal microbiota with periurethral microbiota in GUS. However, there is a study which compares the periurethral and urinary microbiota of women of reproductive age that showed that both environments change after menstruation and intercourse, and as a result, these environments are dynamic and variable like the vaginal microbiota (Price, 2020). Again, urinary, periurethral, vaginal and fecal microbiota were examined in women of reproductive age, urinary microbiota was compared with fecal, and urinary microbiota was shown to be more variable compared with fecal microbiota. However, no comments were made about vaginal and periurethral microbiota in this study (Biehl, 2022). Therefore, our study will be the first to compare these 3 environments in GUS.

Why is periurethral microbiota important?

When we examine the GUS complaints of patients, the situation they describe as pain during intercourse is mainly the pain they feel at the entrance to the vagina, in the introitus. Since this area is close to the skin, we think that bacterial colonization may be different from vaginal colonization. In this patient group, the introitus is generally observed to be more red during examination. This also suggests that aerobic vaginitis agents are more intense in this area. Waetjen has shown in his latest study that there is a density of Streptococcus in the vaginal microbiota of patients with dyspareunia (Waetjen, 2023).

Our hypotheses in this study are: 1-there is a relationship between the vaginal-periurethral and urinary microbiota. 2- Lactobacillus colonization increases in areas outside the vagina with local estrogen treatment. 3- The severity of GUS symptoms is higher in patients with a microbiota predominant by facultative anaerobic bacteria such as Staphylococcus or Streptococcus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been in menopause for at least 1 year
2. Patients with symptoms of genitourinary syndrome (those with symptoms such as vaginal dryness, frequent urination, burning sensation during urination, pain during intercourse)

Exclusion Criteria:

1. Patients with severe overactive bladder symptoms
2. Patients receiving systemic hormone replacement therapy or local estrogen therapy or have received it within the last 3 months
3. Patients using vaginal probiotic products
4. Patients with advanced pelvic organ prolapse
5. Patients with a history of estrogen-dependent breast or endometrial cancer
6. Patients allergic to local estrogen
7. Patients with urinary tract infection at first presentation or patients who have used antibiotics within the last 2 weeks

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Vaginal, periurethral and urinary bladder microbiota | 3 months
  Microbiota contents of 3 areas (vagina, periurethra and bladder) will be obtain and compared to each other

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since this is a human data we cannot share individuals data according to the law but we can share our data as an article

REFERENCES:
- [Background] Mirmonsef P, Hotton AL, Gilbert D, Burgad D, Landay A, Weber KM, Cohen M, Ravel J, Spear GT. Free glycogen in vaginal fluids is associated with Lactobacillus colonization and low vaginal pH. PLoS One. 2014 Jul 17;9(7):e102467. doi: 10.1371/journal.pone.0102467. eCollection 2014. PMID 25033265
- [Background] Mitchell CM, Reed SD, Diem S, Larson JC, Newton KM, Ensrud KE, LaCroix AZ, Caan B, Guthrie KA. Efficacy of Vaginal Estradiol or Vaginal Moisturizer vs Placebo for Treating Postmenopausal Vulvovaginal Symptoms: A Randomized Clinical Trial. JAMA Intern Med. 2018 May 1;178(5):681-690. doi: 10.1001/jamainternmed.2018.0116. PMID 29554173
- [Background] Price TK, Wolff B, Halverson T, Limeira R, Brubaker L, Dong Q, Mueller ER, Wolfe AJ. Temporal Dynamics of the Adult Female Lower Urinary Tract Microbiota. mBio. 2020 Apr 21;11(2):e00475-20. doi: 10.1128/mBio.00475-20. PMID 32317321
- [Background] Ravel J, Brotman RM, Gajer P, Ma B, Nandy M, Fadrosh DW, Sakamoto J, Koenig SS, Fu L, Zhou X, Hickey RJ, Schwebke JR, Forney LJ. Daily temporal dynamics of vaginal microbiota before, during and after episodes of bacterial vaginosis. Microbiome. 2013 Dec 2;1(1):29. doi: 10.1186/2049-2618-1-29. PMID 24451163
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Background] Siddiqui H, Nederbragt AJ, Lagesen K, Jeansson SL, Jakobsen KS. Assessing diversity of the female urine microbiota by high throughput sequencing of 16S rDNA amplicons. BMC Microbiol. 2011 Nov 2;11:244. doi: 10.1186/1471-2180-11-244. PMID 22047020
- [Background] Zhang R, Daroczy K, Xiao B, Yu L, Chen R, Liao Q. Qualitative and semiquantitative analysis of Lactobacillus species in the vaginas of healthy fertile and postmenopausal Chinese women. J Med Microbiol. 2012 May;61(Pt 5):729-739. doi: 10.1099/jmm.0.038687-0. Epub 2012 Feb 2. PMID 22301614
- [Background] Thomas-White K, Taege S, Limeira R, Brincat C, Joyce C, Hilt EE, Mac-Daniel L, Radek KA, Brubaker L, Mueller ER, Wolfe AJ. Vaginal estrogen therapy is associated with increased Lactobacillus in the urine of postmenopausal women with overactive bladder symptoms. Am J Obstet Gynecol. 2020 Nov;223(5):727.e1-727.e11. doi: 10.1016/j.ajog.2020.08.006. Epub 2020 Aug 11. PMID 32791124
- [Background] Waetjen LE, Crawford SL, Gajer P, Brooks MM, Gold EB, Reed BD, Hess R, Ravel J. Relationships between the vaginal microbiota and genitourinary syndrome of menopause symptoms in postmenopausal women: the Study of Women's Health Across the Nation. Menopause. 2023 Nov 1;30(11):1073-1084. doi: 10.1097/GME.0000000000002263. Epub 2023 Oct 2. PMID 37788422
- [Background] The NAMS 2020 GSM Position Statement Editorial Panel. The 2020 genitourinary syndrome of menopause position statement of The North American Menopause Society. Menopause. 2020 Sep;27(9):976-992. doi: 10.1097/GME.0000000000001609. PMID 32852449
- [Background] Lillemon JN, Karstens L, Nardos R, Garg B, Boniface ER, Gregory WT. The Impact of Local Estrogen on the Urogenital Microbiome in Genitourinary Syndrome of Menopause: A Randomized-Controlled Trial. Female Pelvic Med Reconstr Surg. 2022 Jun 1;28(6):e157-e162. doi: 10.1097/SPV.0000000000001170. Epub 2022 Apr 15. PMID 35420551
- [Background] Brotman RM, Shardell MD, Gajer P, Fadrosh D, Chang K, Silver MI, Viscidi RP, Burke AE, Ravel J, Gravitt PE. Association between the vaginal microbiota, menopause status, and signs of vulvovaginal atrophy. Menopause. 2014 May;21(5):450-8. doi: 10.1097/GME.0b013e3182a4690b. PMID 24080849
- [Background] Biehl LM, Farowski F, Hilpert C, Nowag A, Kretzschmar A, Jazmati N, Tsakmaklis A, Wieters I, Khodamoradi Y, Wisplinghoff H, Vehreschild MJGT. Longitudinal variability in the urinary microbiota of healthy premenopausal women and the relation to neighboring microbial communities: A pilot study. PLoS One. 2022 Jan 14;17(1):e0262095. doi: 10.1371/journal.pone.0262095. eCollection 2022. PMID 35030190
- [Background] Anglim B, Phillips C, Shynlova O, Alarab M. The effect of local estrogen therapy on the urinary microbiome composition of postmenopausal women with and without recurrent urinary tract infections. Int Urogynecol J. 2022 Aug;33(8):2107-2117. doi: 10.1007/s00192-021-04832-9. Epub 2021 May 18. PMID 34003309